CLINICAL TRIAL: NCT05072912
Title: Screening Study to Identify Patients With Complement Factor I Deficiencies
Status: Terminated | Type: Observational
Why Stopped: Enrollment
Sponsor: Catalyst Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: CFI-001
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Previous Diagnosis With a Complement-mediated Disease and/or With Clinical Manifestations Reasonably Associated With Complement Factor I Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is screening study to identify patients with Complement Factor I deficiencies. The primary objective is to identify participants with CFI deficiencies and assess the prevalence in the screened population.

ELIGIBILITY:
Inclusion Criteria:

An individual must meet all the following criteria to be eligible to participate in this study:

1. A male or female ≥6 months of age who has been diagnosed with a complement-mediated disease in which a reasonable etiological association with CFI deficiency has been reported
2. Affirmation of participant's informed consent or LAR's willingness to provide informed consent with signature confirmation before any study-related activities. (Study-related activities are any procedures that would not have been performed during normal clinical management of the participant.) The participant (if a minor) must be willing to give written informed assent if the minor is within the age groups 7 to 11 years old and 12 to 17 years old.

Exclusion Criteria:

1) Diagnosis of age-related macular degeneration that is complement-related with no concurrent systemic complement involvement

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients previously diagnosed with a complement-mediated disease and/or with clinical manifestations in which a reasonable etiological association with Complement Factor I (CFI) deficiency has been reported.
  Examples of these diseases and conditions are (but not limited to): atypical hemolytic uremic syndrome, Complement 3 Glomerulopathy, membranoproliferative glomerulonephritis, systemic lupus erythematosus, leukocytoclastic vasculitis, recurrent bacterial infections, unexplained inflammation or edema, and some autoimmune disorders.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Complement Factor I Deficiency Identification | At Screening
  Identification of participants with a CFI deficiency and percentage of those with a CFI deficiency versus total number of screened participants

SECONDARY OUTCOMES:
Demographics, Disease Characteristics, Medication Use | At Screening
  Demographics, disease characteristics (including disease history), and disease-related medication use. Complement levels and mutation data will also be collected from medical records, if previously assessed and available.

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Consultants, LLC, Huntsville, Alabama, United States